CLINICAL TRIAL: NCT03493139
Title: Physical Activity Across the Curriculum (PAAC 3):Teacher vs. Remotely Delivered Classroom Physical Activity Breaks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00141841; R01DK085317 (NIH)
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2020-09

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Classroom Physical Activity Breaks Delivered by Teacher vs. Classroom Physical Activity Breaks Delivered by Video
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAAC-R (Experimental): Physical Activity Across the Curriculum-Remote (PAAC-R) will include protocol specific activity breaks delivered remotely via a television in the classroom.
  Interventions: Behavioral: Physical Activity Across the Curriculum
- PAAC-T (Experimental): Physical Activity Across the Curriculum-Teacher (PAAC-T) will include protocol specific activity breaks delivered by the classroom teacher.
  Interventions: Behavioral: Physical Activity Across the Curriculum

INTERVENTIONS:
Behavioral: Physical Activity Across the Curriculum — Activity breaks will be designed for delivery in the classroom without reconfiguration of the classroom space. Activities will emphasize whole body movements, using large muscle groups. Each break includes multiple activities. Each activity lasts about 2 minutes. There will be a total of about 20 minutes of physical activity done each school day.

SUMMARY:
The study is designed to compare two methods of delivering short (~10 min) physical activity breaks that will occur during the regular school day for 3 years. Schools will be randomized to deliver physical activity breaks led by either the regular classroom teacher or by a remote instructor through a video in the classroom. Both delivery methods will promote a variety of whole body movements using large muscle groups. The schools will not be able to choose which group (regular teacher or remote instructor) they will be part of.

ELIGIBILITY:
Inclusion Criteria:

* 2nd and 3rd grade students

Exclusion Criteria:

* Students who are confined to a wheel chair, blind, or intellectually disadvantaged may be unable perform tests for cardiovascular fitness or MVPA using accelerometers

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 470 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Moderate-to-vigorous physical activity (MVPA) time during activity breaks | Year 3
  Measure will be calculated as the average number of minutes of moderate to vigorous physical activity (MVPA) during the period of activity breaks. Measure will be captured using an accelerometer.

SECONDARY OUTCOMES:
MVPA time during the school day | Year 3
  Measure will be calculated as the average number of minutes of moderate to vigorous physical activity (MVPA) during the school day. Measure will be captured using an accelerometer.
Total daily MVPA | Year 3
  Measure will be calculated as the average number of minutes of moderate to vigorous physical activity (MVPA) during the entire day. Measure will be captured using an accelerometer.
Body mass index (BMI) | Fall Semester Year 1
  Weight and height will be combined to report BMI in kg/m^2.
Body mass index (BMI) | Spring Semester Year 1
  Weight and height will be combined to report BMI in kg/m^2.
Body mass index (BMI) | Spring Semester Year 2
  Weight and height will be combined to report BMI in kg/m^2.
Body mass index (BMI) | Spring Semester Year 3
  Weight and height will be combined to report BMI in kg/m^2.
Energy expenditure of activity breaks | Year 2
  Calculated as the number of calories used during a classroom activity break.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Donnelly, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
Please contact PI.
Supporting Information: Study Protocol
Time Frame: After 1/2026

REFERENCES:
- [Background] Szabo-Reed AN, Washburn RA, Greene JL, Ptomey LT, Gorczyca A, Lee RH, Little TD, Lee J, Honas J, Donnelly JE. Physical activity across the curriculum (PAAC3): Testing the application of technology delivered classroom physical activity breaks. Contemp Clin Trials. 2020 Mar;90:105952. doi: 10.1016/j.cct.2020.105952. Epub 2020 Jan 29. PMID 32006633